CLINICAL TRIAL: NCT01555372
Title: Treatment of Unstable Distal Clavicular Fractures (Neer 2b): Hook Plate vs Locking Plate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Nanjing Medical University (Other); The First People's Hospital of Huzhou (Other); Huai'an No. 2 People's Hospital (Unknown); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Leisheng Jiang, director of department of Orthopaedic,Xinhua hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U2032001
Record Dates: First submitted 2012-03-11; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Clavicle Injuries
Keywords: unstable distal clavicular fractures (Neer 2b); Study Protocol; Fracture Fixation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hook Plate (Active Comparator): 20 participants will be enrolled in this group.
  Interventions: Device: Hook Plate
- Locking Plates (Experimental): 20 paticipants will be enrolled in this group
  Interventions: Device: Locking Plate

INTERVENTIONS:
Device: Hook Plate — All participants will have an open reduction internal fixation. The affected upper limb will be temporarily fixed by a sling after admission. Under necessary test, general anaesthetic and antibiotic prophylaxis, the patients will be placed in a beach-chair position in an orthopaedic theatre. The operated side will be prepped and draped and a transverse incision will be made over the fracture site. The fracture ends will be identified, reduced and fixed with HP. X-ray was applied to check the grade of reduction before the operation is completed. Post-operative care will include early active mobilization managed by a standard physiotherapy rehabilitation regime.
  Arms: Hook Plate
Device: Locking Plate — All participants will have an open reduction internal fixation. The affected upper limb will be temporarily fixed by a sling after admission. Under necessary test, general anaesthetic and antibiotic prophylaxis, the patients will be placed in a beach-chair position in an orthopaedic theatre. The operated side will be prepped and draped and a transverse incision will be made over the fracture site. The fracture ends will be identified, reduced and fixed with locking plate. X-ray was applied to check the grade of reduction before the operation is completed. Post-operative care will include early active mobilization managed by a standard physiotherapy rehabilitation regime.
  Arms: Locking Plates

SUMMARY:
The investigators propose to test the hypotheses that compared with Hook Plate (HP), Locking Plate (LP) reduces the postoperative complications and leads to a better functional recovery after unstable distal clavicle fractures (Neer 2b).

DETAILED DESCRIPTION:
Controversy exists regarding the optimal treatment for patients with unstable distal clavicular fractures (Neer 2b). The recognized treatment alternatives are Hook plate.Notably, criticisms on this fixation method also appeared and the potential risks of hook migration, loosening, subacromial impingement or rotator cuff injury, and acromial osteolysis were still unsolved. Recently, Herrmann et al.and Largo et al.stabilized the distal clavicle with Locking plate (LP) and these studies offered encouraging support for LP. Because of small sample size (27 patients) and nonrandomization, the convictive power of these researches is not strong enough.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Unstable fractures of distal clavicle (Neer 2b fractures), acute or chronic and unilateral fractures.
3. Normal shoulder functions before injury.
4. Internal fixation with either HP or LP.
5. The subjects were in good health and were able to comply with all prescribed follow-up procedures.

Exclusion Criteria:

1. Patients who present multiple traumas.
2. Patients with other serious injuries to either upper limb that would interfere with rehabilitation.
3. Patients with a pathological, recurrent or open clavicle fracture.
4. Patient unwilling to give written informed consent.
5. Patients with cognitive impairment unable to comply with treatment programme.
6. Patients with a serious disorder of bone metabolism other than osteoporosis (e.g., endocrine bone diseases, osteomalacia and Paget's disease)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
the postoperative complications | 12 months
  complication that related with surgery or fracture will be defined as any event that necessitated another operative procedure or additional medical treatment

SECONDARY OUTCOMES:
the affected limb function | 3, 6, 9,12 months
  the affected limb function measured using the Constant-Murley Score and using the Disabilities of the Arm, Shoulder and Hand (DASH) Score measured at 3, 6,9and 12months post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng L Jiang, doctor, Study Chair — Orthopaedic department, Shanghai Jiaotong University Xinhua Hospital
Locations (1):
- Orthopaedic department,Xinhua hospital affiliated to Shanghai JiaoTong University School of Medicine, Shanghai, China